CLINICAL TRIAL: NCT03069963
Title: A Randomized, Open Label, 2-Treatment Crossover Study to Compare by pH Metry, the Antacid Activity of the To-be-registered Product (250 mg Sodium Alginate/187.5 mg Calcium Carbonate/106.5 mg Sodium Hydrogen Carbonate, Chewable Tablets) Versus the Registered Gaviscon Double Action Tablets, in Healthy Adult Subject
Brief Title: PH Metry Study to Compare the Antacid Activity of Z0063 Versus Gaviscon Double Action Tablets, in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PDY14362; 2015-000763-13 (EudraCT Number); U1111-1183-5042 (Other: UTN)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2017-06

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — alginate, aluminium hydroxide, magnesium trisilicate, sodium bicarbonate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Z0063 to Gaviscon) (Experimental): The subjects will be given Z0063 single dose and then will crossover to Gaviscon single dose
  Interventions: Drug: Z0063; Drug: Gaviscon
- Sequence 2 (Gaviscon to Z0063) (Experimental): The subjects will be given Gaviscon single dose and then will crossover to Z0063 single dose
  Interventions: Drug: Z0063; Drug: Gaviscon

INTERVENTIONS:
Drug: Z0063 — Pharmaceutical form: chewable tablets
  Route of administration: oral
Drug: Gaviscon — Pharmaceutical form: chewable tablets
  Route of administration: oral

SUMMARY:
Primary Objective:

Pharmacodynamics: assessment by pH metry of the change in gastric pH (antacid activity) of Z0063, in comparison to the effect of Gaviscon Double Action Tablets, in healthy adult subjects.

Secondary Objective:

Safety: assessment of the clinical safety of Z0063, and Gaviscon Double Action Tablets, in healthy adult subjects.

DETAILED DESCRIPTION:
The maximal total study duration per subject is 5 weeks and 1 day.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 55 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 28.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs, electrocardiogram (ECG) and laboratory parameters.
* Subject has to accept a gastric probe.

Exclusion criteria:

* Any history or presence of clinically relevant abnormalities at screening which could interfere with the objectives of the study or the safety of the subject's participation.
* Blood donation, any volume, within 2 months before inclusion.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* If female, pregnancy (defined as positive beta-human chorionic gonadotropin [β-HCG] blood test), breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Any subject in the exclusion period of a previous study according to applicable regulations.
* Any subject who cannot be contacted in case of emergency.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
* Positive result on urine drug screen.
* Positive alcohol breath test.
* Known hypersensitive to alginates, products or formulation excipients, and/or to any component of the standardized meal.
* Any subject with difficulty in chewing and swallowing.
* Any subject with strong gag reflex.
* Any intake of aluminium and magnesium containing antacids or other alginate-containing medicinal products within 14 days before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-04-23 (Actual); Study Completion 2017-04-23 (Actual)

PRIMARY OUTCOMES:
Percentage of time at which the intragastric pH is at least equal to or greater than 4 during the 4-hour observation period post-dose | 4 hours after the investigational medicinal product (IMP) administration

SECONDARY OUTCOMES:
Percentage of time at which the intragastric pH is at least equal to or greater than 3 during the 4-hour observation period post-dose | 4 hours after the IMP administration
4-hour median pH | 4 hours after the IMP administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 2500001, Gières, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org